CLINICAL TRIAL: NCT01706965
Title: 6R-BH 4 in People With Schizophrenia and Schizoaffective Disorder
Brief Title: Kuvan in People With Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6320
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — sapropterin; Geritol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kuvan (Experimental): Kuvan once-daily dosing initiated with 10mg/kg for the first week followed by 20mg/kg for the remaining weeks of the study
  Interventions: Drug: Kuvan
- Multivitamin (Active Comparator): Daily multivitamin tablet
  Interventions: Drug: Multivitamin

INTERVENTIONS:
Drug: Kuvan — 20mg/kg using a daily dosing schedule. To increase tolerability, treatment will be initiated at 10mg/kg for the first week of the study. Given the short length of the trial, no dose adjustments will be made for changes in weight
  Other Names: Sapropterin dihydrochloride
  Arms: Kuvan
Drug: Multivitamin — Multi-vitamin will be used as an active control in this study. Will be dosed daily
  Arms: Multivitamin

SUMMARY:
Rater blinded trial of six weeks of Kuvan vs. multivitamin in 60 outpatients with schizophrenia or schizoaffective disorder. The aims are to evaluate an anticipated clinical response to Kuvan treatment including negative symptom and cognitive deficits, evaluate safety of Kuvan treatment for schizophrenic patients and evaluate the relationship of changes in plasma Kuvan levels and efficacy outcomes.

DETAILED DESCRIPTION:
Tetrahydrobiopterin (BH4) is a vital central nervous system (CNS) cofactor that maintains availability of amine neurotransmitters such as dopamine (DA) and serotonin (5HT), and stimulates and modulates the glutamatergic system. Dysregulation of these neurotransmitter systems has been implicated in the pathogenesis of schizophrenia (SZ). A central role of BH4 in schizophrenia is further supported by a study finding a relative deficit of 32% for SZ patients as compared to controls. The observed BH4 deficit is comparable to that reported for genetic BH4 deficiency disorders, supporting its characterization as having physiological significance. This highly significant finding, along with: a) the known roles of BH4 in neurotransmitter maintenance, b) dysregulation of CNS neurotransmitter synthesis observed in human BH4 deficiencies, c) evidence that plasma biopterin levels are correlated with CNS biopterin levels, and d) evidence that urinary biopterin excretion is not increased in SZ, all support our hypothesis that dysregulation of BH4 biosynthesis is involved in the pathophysiology of SZ. Moreover, additional data suggesting that mood stabilizer drugs can moderately increase levels of biopterin in patients with psychiatric disorders, and the reported efficacy of BH4 in pilot studies of neuropsychiatric disorders, suggest that alleviation of the schizophrenia BH4 deficit via treatment with synthetic BH4 supplement (Sapropterin dihydrochloride or Kuvan), may give rise to an improvement of the symptoms of schizophrenia, including positive and negative symptoms as well as neurocognitive deficits. Sapropterin dihydrochlorides, teh active pharmaceutical ingredient in Kuvan Tablets,is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4)

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients with schizophrenia or schizoaffective disorder
* Ages 18-64
* A score of 45 or greater on PANSS
* All oral and depot antipsychotics (with the exception of clozapine) are allowable. Patients must be on their antipsychotic medication for 3 months and stable on dose of antipsychotic and adjunctive medications for 2 weeks prior to study entry. If a patient is on depot medication, they must be stable in dose for 2 months

Exclusion Criteria:

* Organic brain disorder, including epilepsy; mental retardation; or a medical condition whose pathology or treatment would likely alter the presentation or treatment of schizophrenia
* Participated in any investigational study or taken an investigational drug within 30 days
* Current Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) diagnosis of drug/alcohol abuse in last month and current DSM-IV diagnosis drug/alcohol dependence in last 6 months. Subjects must have a negative drug screen at baseline (with one retest allowed for suspected false positive based on clinical judgement of the investigator)
* Diagnosis of any known BH4 deficiency disorder (other than schizophrenia or schizoaffective disorder), including dopa-responsive dystonia,phenylketonuria (PKU), and autism
* Current treatment with clozapine
* In the investigator's judgment, a significant risk of suicide or violent behavior
* Current use of levodopa and nitric oxide-mediated vasorelaxation or oral minoxidil
* Women will be excluded if they are pregnant, lactating, or not either surgically-sterile or using appropriate methods of birth control. Women must agree to continue using applicable birth control throughout the trial. All women of child-bearing potential must have a negative urine pregnancy test at the screening visit and visit 2 (1 week before beginning study medication)
* Absolute neutrophil count below 2.0 on screening
* Any contraindication or allergic reaction to previous multi-vitamin or unwillingness to stop use of current multi-vitamin during study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, M.D., Principal Investigator — New York State Psychiatric
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kuvan | Multivitamin
Started | 14 | 13
Completed | 13 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kuvan | Multivitamin | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.15 (12.1) | 46.1 (8.0) | 43.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 3 | 6 | 9
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Final Positive and Negative Symptom Scale (PANSS)
Description: This is a is a 30 item rating scale widely used in the assessment of schizophrenia ranging from 30-210. Higher scores are worse
Time Frame: Baseline (start of Kuvan) and at six weeks of treatment
Measure: Mean (Standard Deviation); unit: PANSS Total
Arm/Group | Kuvan | Multivitamin
Number analyzed (Participants) | 13 | 12
PANSS Total | 54.4 (10.9) | 60.2 (13.7)
Statistical Analysis 1: Comparison: Kuvan vs Multivitamin; Univariate ANOVA, controlling for baseline PANSS total; Test type: Superiority; p = .38, ANOVA

2. Primary Outcome: Final MATRICS Cognitive Battery
Description: MATRICS assessing 7 domains (Speed of Processing, Attention/Vigilance, Working Memory, Verbal Learning, Visual Learning, Reasoning and Problem Solving, and Social Cognition. Raw scores are converted into a composite T-score (normative mean = 50; standard deviation = 10), where higher values indicated less impairment.
Time Frame: Baseline to week 6
Measure: Mean (Standard Deviation); unit: Total MATRICS score
Arm/Group | Kuvan | Multivitamin
Number analyzed (Participants) | 13 | 12
Total MATRICS score | 33.92 (17.1) | 35.0 (12.5)
Statistical Analysis 1: Comparison: Kuvan vs Multivitamin; Test type: Superiority — ANOVA, controlled for baseline MATRICS; p = .99, ANOVA

ADVERSE EVENTS:
Arm/Group | Kuvan | Multivitamin
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 8/13 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kuvan (N=13) | Multivitamin (N=12)
constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dizziness (General disorders) | 4 (4) | 1 (1)
nocturnal enuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stomach disconfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
restlessnes (Psychiatric disorders) | 1 (1) | 2 (2)
stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
URI (Infections and infestations) | 1 (1) | 0 (0)
Difficulty speaking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
headache (Gastrointestinal disorders) | 0 (0) | 2 (2)
urtiacia (Immune system disorders) | 0 (0) | 1 (1)
Vaginal Yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
auditory hallucinatiuons (Psychiatric disorders) | 0 (0) | 1 (1)
anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No